CLINICAL TRIAL: NCT01754103
Title: Neuroplasticity in Blind Subjects After Repetitive Tactile Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Tomas Ortiz Alonso, MD PhD, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: VISION TACTIL
Record Dates: First submitted 2012-07-02; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Blindness
Keywords: blind; tactile stimulation; cross-modality; visual qualia; resting state MRI; functional connectivity; neuroplasticity
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Connectivity MRI (Experimental): Functional Connectivity will be measured by MRI, we will perform one T1WI run as well as three resting state bold based runs. Bold runs parameters: TE 30ms, TR 3000ms, flip angle 90º, gap 0mm, 124 time points, voxel size 3mm, duration 6min18s each, FOV 240x240x141.
  Interventions: Other: Tactile Training

INTERVENTIONS:
Other: Tactile Training — Tactile Training to induce neuroplasticity in the visual pathway, measured with functional connectivity MRI

SUMMARY:
Brain plasticity of cortical activity caused by repetitive tactile stimulation could have a progressive development that was from primary parietal areas, passing over parieto-occipital areas and came secondary to primary occipital areas. This process allows to understand the existence of neurons in the brain and specific areas for certain functions independent of the type of stimulation is performed.

By performing repetitive tactile stimulation over a period of 3 months,using a tactile stimulator, our group will try to prove several that repetitive tactile stimulation can create cross-modality and improve recognition and localization of patterns in blind people.

DETAILED DESCRIPTION:
The investigators will use passive repetitive tactile stimulation over a period of 3 months, one hour a day for five days a week, with vertical, horizontal and oblique lines generated randomly by a tactile stimulator. Our aim is (a) to study if repetitive tactile stimulation can create cross-modality and improve recognition and localization of patterns in blind people, (b) to evaluate the impact of this training on brain activity the investigators performed high-density scalp EEG recording during the initial stimulation session and in the last one. And (c) measure the functional connectivity of the brain with resting state MRI pre and post training. The resting state MRI protocol consist on one run of T1WI and three bold runs (TE=30ms,TR=3000ms, flip angle 90º,voxel size 3mm, 124 time points, 0 gap).

Cross-modality sensory stimulation may offer a good opportunity to improve recognition, localization and navigation in blind people. Although the neural substrate of this multimodality integration is not fully understood yet. Some areas of the brain, mainly the lateral occipital cortex, are specialized for visual object recognition and they can be activated by tactile stimuli. This activation of the visual cortex might lead to visual-like perception, regardless of the sensory input modality.

In the blind the high demand required by object recognition appears to recruit also ventral and dorsal occipital areas. Blindness modifies neocortical processing of non-visual tasks, including frontoparietal and visual regions during tactile stimulation. It is also known that people with blindness proficient in the use of a visuo-tactile sensory substitution device that presents visual images as patterns of electric stimuli to the subject's tongue, like Bach-y-Rita and Ptito said, show occipital cortex activation in an orientation-discrimination task.

As far as the investigators know there are no studies aimed at understanding the relationship between activation of lateral occipital cortex and the ability to recognize objects presented to the hand along time. In particular, the investigators tested if repetitive passive tactile stimulation leads to activation of visual areas and recognition of spatial patterns in people with blindness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis: Different Causes of blindness were diverse: congenital nystagmus, glaucoma, retinopathy, congenital cataracts, lenticular fibroplasia, macular degeneration, optic atrophy, Peter's anomaly with microphthalmia, retinal detachment, retina necrosis, retinitis pigmentosa and uveitis

Exclusion Criteria:

* No history of neurological, psychiatric, cognitive or sensorimotor deficits other than blindness.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
MRI Functional Connectivity of the visual pathway | 1 year
  Functional Connectivity analysis (fcMRI) is a tool that allows functionally associated brain regions to be identified. fcMRI takes advantage of the observation that the brain regions exhibit spontaneous, low frequency variations as measured using blood oxygenation level-dependent (BOLD) imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Tomás Ortiz Alonso, MD PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Pascual-Leone A, Amedi A, Fregni F, Merabet LB. The plastic human brain cortex. Annu Rev Neurosci. 2005;28:377-401. doi: 10.1146/annurev.neuro.27.070203.144216. PMID 16022601
- [Background] Feldman DE, Brecht M. Map plasticity in somatosensory cortex. Science. 2005 Nov 4;310(5749):810-5. doi: 10.1126/science.1115807. PMID 16272113
- [Background] van Praag H, Christie BR, Sejnowski TJ, Gage FH. Running enhances neurogenesis, learning, and long-term potentiation in mice. Proc Natl Acad Sci U S A. 1999 Nov 9;96(23):13427-31. doi: 10.1073/pnas.96.23.13427. PMID 10557337
- [Background] Greenwood RS, Parent JM. Damage control: the influence of environment on recovery from brain injury. Neurology. 2002 Nov 12;59(9):1302-3. doi: 10.1212/wnl.59.9.1302. No abstract available. PMID 12427874
- [Background] Lepore N, Voss P, Lepore F, Chou YY, Fortin M, Gougoux F, Lee AD, Brun C, Lassonde M, Madsen SK, Toga AW, Thompson PM. Brain structure changes visualized in early- and late-onset blind subjects. Neuroimage. 2010 Jan 1;49(1):134-40. doi: 10.1016/j.neuroimage.2009.07.048. Epub 2009 Jul 28. PMID 19643183
- [Background] Elbert T, Sterr A, Rockstroh B, Pantev C, Muller MM, Taub E. Expansion of the tonotopic area in the auditory cortex of the blind. J Neurosci. 2002 Nov 15;22(22):9941-4. doi: 10.1523/JNEUROSCI.22-22-09941.2002. PMID 12427851
- [Background] Fortin M, Voss P, Lord C, Lassonde M, Pruessner J, Saint-Amour D, Rainville C, Lepore F. Wayfinding in the blind: larger hippocampal volume and supranormal spatial navigation. Brain. 2008 Nov;131(Pt 11):2995-3005. doi: 10.1093/brain/awn250. Epub 2008 Oct 14. PMID 18854327
- [Background] Sadato N, Pascual-Leone A, Grafman J, Ibanez V, Deiber MP, Dold G, Hallett M. Activation of the primary visual cortex by Braille reading in blind subjects. Nature. 1996 Apr 11;380(6574):526-8. doi: 10.1038/380526a0. PMID 8606771
- [Background] Sadato N, Pascual-Leone A, Grafman J, Deiber MP, Ibanez V, Hallett M. Neural networks for Braille reading by the blind. Brain. 1998 Jul;121 ( Pt 7):1213-29. doi: 10.1093/brain/121.7.1213. PMID 9679774
- [Background] Merabet LB, Hamilton R, Schlaug G, Swisher JD, Kiriakopoulos ET, Pitskel NB, Kauffman T, Pascual-Leone A. Rapid and reversible recruitment of early visual cortex for touch. PLoS One. 2008 Aug 27;3(8):e3046. doi: 10.1371/journal.pone.0003046. PMID 18728773
- [Background] Burton H, Sinclair RJ, McLaren DG. Cortical activity to vibrotactile stimulation: an fMRI study in blind and sighted individuals. Hum Brain Mapp. 2004 Dec;23(4):210-28. doi: 10.1002/hbm.20064. PMID 15449356
- [Background] Wheat HE, Goodwin AW, Browning AS. Tactile resolution: peripheral neural mechanisms underlying the human capacity to determine positions of objects contacting the fingerpad. J Neurosci. 1995 Aug;15(8):5582-95. doi: 10.1523/JNEUROSCI.15-08-05582.1995. PMID 7643203
- [Background] Amedi A, Stern WM, Camprodon JA, Bermpohl F, Merabet L, Rotman S, Hemond C, Meijer P, Pascual-Leone A. Shape conveyed by visual-to-auditory sensory substitution activates the lateral occipital complex. Nat Neurosci. 2007 Jun;10(6):687-9. doi: 10.1038/nn1912. Epub 2007 May 21. PMID 17515898
- [Background] Swisher JD, Halko MA, Merabet LB, McMains SA, Somers DC. Visual topography of human intraparietal sulcus. J Neurosci. 2007 May 16;27(20):5326-37. doi: 10.1523/JNEUROSCI.0991-07.2007. PMID 17507555
- [Background] Harris JA, Miniussi C, Harris IM, Diamond ME. Transient storage of a tactile memory trace in primary somatosensory cortex. J Neurosci. 2002 Oct 1;22(19):8720-5. doi: 10.1523/JNEUROSCI.22-19-08720.2002. PMID 12351747
- [Background] De Volder AG, Catalan-Ahumada M, Robert A, Bol A, Labar D, Coppens A, Michel C, Veraart C. Changes in occipital cortex activity in early blind humans using a sensory substitution device. Brain Res. 1999 Apr 24;826(1):128-34. doi: 10.1016/s0006-8993(99)01275-5. PMID 10216204
- [Background] Gizewski ER, Gasser T, de Greiff A, Boehm A, Forsting M. Cross-modal plasticity for sensory and motor activation patterns in blind subjects. Neuroimage. 2003 Jul;19(3):968-75. doi: 10.1016/s1053-8119(03)00114-9. PMID 12880825
- [Background] Zarei M, Johansen-Berg H, Smith S, Ciccarelli O, Thompson AJ, Matthews PM. Functional anatomy of interhemispheric cortical connections in the human brain. J Anat. 2006 Sep;209(3):311-20. doi: 10.1111/j.1469-7580.2006.00615.x. PMID 16928200
- [Background] Hofer S, Frahm J. Topography of the human corpus callosum revisited--comprehensive fiber tractography using diffusion tensor magnetic resonance imaging. Neuroimage. 2006 Sep;32(3):989-94. doi: 10.1016/j.neuroimage.2006.05.044. Epub 2006 Jul 18. PMID 16854598
- [Background] Mahncke HW, Connor BB, Appelman J, Ahsanuddin ON, Hardy JL, Wood RA, Joyce NM, Boniske T, Atkins SM, Merzenich MM. Memory enhancement in healthy older adults using a brain plasticity-based training program: a randomized, controlled study. Proc Natl Acad Sci U S A. 2006 Aug 15;103(33):12523-8. doi: 10.1073/pnas.0605194103. Epub 2006 Aug 3. PMID 16888038
- [Background] Karni A, Meyer G, Jezzard P, Adams MM, Turner R, Ungerleider LG. Functional MRI evidence for adult motor cortex plasticity during motor skill learning. Nature. 1995 Sep 14;377(6545):155-8. doi: 10.1038/377155a0. PMID 7675082
- [Background] Gougoux F, Zatorre RJ, Lassonde M, Voss P, Lepore F. A functional neuroimaging study of sound localization: visual cortex activity predicts performance in early-blind individuals. PLoS Biol. 2005 Feb;3(2):e27. doi: 10.1371/journal.pbio.0030027. Epub 2005 Jan 25. PMID 15678166